CLINICAL TRIAL: NCT05039905
Title: Development of the Surgical Technique Using Radioactive Fluorescent Dual Contrast Agent for Intraoperative Sentinel Lymph Node Detection in Lung Cancer Patients
Brief Title: SLN Detection With Tc-MSA-ICG in Lung Cancer Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor of Thoracic and Cardiovascular Surgery, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020GR0436
Record Dates: First submitted 2021-02-15; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Sentinel lymph node; Radioactive fluorescent dual contrast agent
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Lung cancer patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-MSA-ICG injection (Experimental): 99mTc-MSA-ICG injection
  1mCi of 99mTc
  1mg of MSA 0.1mg of ICG Total 1cc injection volume at 2 hours before the surgery
  Interventions: Drug: 99mTc-MSA-ICG

INTERVENTIONS:
Drug: 99mTc-MSA-ICG — Intratumoral injection of 99mTechnetium-manosylated albumin-indocyanine green to lung cancer patients

SUMMARY:
It is necessary to develop a technique of sentinel lymph node detection using radioactive fluorescent dual contrast agent consisting targetable albumin for specific marker to accurately determine whether or not the sentinel lymph nodes have metastasized or non-metastasized. Therefore, investigators would like to conduct a clinical trial to evaluate the effectiveness of radioactive fluorescent dual contrast agent to detect sentinel lymph nodes for patient-specific minimally invasive surgery.

DETAILED DESCRIPTION:
It is necessary to develop a technique of sentinel lymph node detection using radioactive fluorescent dual contrast agent consisting targetable albumin for specific marker to accurately determine whether or not the sentinel lymph nodes have metastasized or non-metastasized. Therefore, investigators would like to conduct a clinical trial to evaluate the effectiveness of radioactive fluorescent dual contrast agent (99mTc-MSA-ICG) to detect sentinel lymph nodes for patient-specific minimally invasive surgery.

To analyze the effectiveness of radioactive fluorescent dual contrast agent (99mTc-MSA-ICG) for detecting sentinel lymph node, total 10 lung cancer patients will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

Preoperative examinations (chest CT, PET/CT, bone scan, brain MRI) diagnosed the clinical stage as T1a or T1b with the size the cancer less than 2 cm and adenocarcinoma or square cell carcinoma through preoperative biopsy, with no lymph node or other diseases and lung disease. A person who meets the conditions described below and does not fall under the exclusion criteria is selected as an adult.

* Eastern cooperative oncology group (ECOG) performance scale: 0~2
* White blood cell count ≥ 3,000/㎣ and ≤ 12,000/㎣
* Neutrophil count ≥ 1,500/㎣
* Platelet count ≥ 100,000/㎣
* AST, ALT ≤ 2.5 times the upper limit
* Total bilirubin ≤ 2.5 times the upper limit
* Serum creatinine ≤ 1.5 time the upper limit

Exclusion Criteria:

* Those who do not agree or refuse to participate in the research
* A person who is not suitable for general anesthesia
* A person with a clinically significant acute or unstable condition
* A person with the following serious heart disease

  1. congestive heart failure with symptoms
  2. New York Heart Association III/IV Class Heart Disease
  3. Unstable angina
  4. Symptom or unregulated heart arrhythmia
  5. Myocardial infarction within the past three months
  6. QT interval (QTcF) using Fridricia calibration
  7. Family history of long QT syndrome
* Those who cannot be scanned (e.g., patients with claustrophobia, ect.)
* A person who received a therapeutic radiation dose within four weeks prior to participation in the study ([18F]FDG has a half-life of 109 minutes, so after 18.2 hours, 99mTc-MDP has a half-life of 6 hours, that is after 2.5 days)
* A person who is being administered drugs such as a drug metabolic enzyme inducer or inhibitor within four weeks before participating in the study
* A person who has overreacted or had side effects on clinical research medications (ICG or 99mTc).
* Patients with closed diseases
* Patients with iodine intolerance
* In the case of pregnant women/feeding mothers or pregnant women, those who do not agree to the use of appropriate contraception methods during the research period;
* A person who participated in another clinical study within 12 weeks before participating in the study and administered clinical research medications or received medical device procedures for clinical research.
* Those who are unfit to participate in this clinical study in the judgment of the research manager

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical chemistry examination-1 (CRP,Cholesterol,Ca,total,TotalBilirubin,directBilirubin,BUN,Creatinine,Phosphorus, inorganic) | Within two weeks before surgery
  Carrying out the clinical chemistry examination(CRP,Cholesterol,Ca,total,TotalBilirubin,directBilirubin,BUN,Creatinine,Phosphorus, inorganic) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery. (mg/dL)
Clinical chemistry examination-2 | postoperative day 0
  Carrying out the clinical chemistry examination(CRP,Cholesterol,Ca,total,TotalBilirubin,directBilirubin,BUN,Creatinine,Phosphorus, inorganic) to check the drug-related safety in 10 lung cancer patients on postoperativeday(POD) 0 (mg/dL)
Clinical chemistry examination-3 | postoperative day 1
  Carrying out the clinical chemistry examination(CRP,Cholesterol,Ca,total,TotalBilirubin,directBilirubin,BUN,Creatinine,Phosphorus, inorganic) to check the drug-related safety in 10 lung cancer patients on POD 1 (mg/dL)
Clinical chemistry examination-4 | postoperative day 5
  Carrying out the clinical chemistry examination(CRP,Cholesterol,Ca,total,TotalBilirubin,directBilirubin,BUN,Creatinine,Phosphorus, inorganic) to check the drug-related safety in 10 lung cancer patients on POD 5 (mg/dL)
Clinical chemistry examination-5 | within two weeks before surgery
  Carrying out the clinical chemistry examination (Procalcitonin) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery. (ng/mL)
Clinical chemistry examination-6 | postoperative day 0
  Carrying out the clinical chemistry examination (Procalcitonin) to check the drug-related safety in 10 lung cancer patients on POD 0 (ng/mL)
Clinical chemistry examination-7 | postoperative day 1
  Carrying out the clinical chemistry examination (Procalcitonin) to check the drug-related safety in 10 lung cancer patients on POD 1 (ng/mL)
Clinical chemistry examination-8 | postoperative day 5
  Carrying out the clinical chemistry examination (Procalcitonin) to check the drug-related safety in 10 lung cancer patients on POD 5 (ng/mL)
Clinical chemistry examination-9 | within two weeks before surgery
  Carrying out the clinical chemistry examination (AST,ALT,LDH,ALP,GGT) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (IU/L)
Clinical chemistry examination-10 | postoperative day 0
  Carrying out the clinical chemistry examination (AST,ALT,LDH,ALP,GGT) to check the drug-related safety in 10 lung cancer patients on POD 0 (IU/L)
Clinical chemistry examination-11 | postoperative day 1
  Carrying out the clinical chemistry examination (AST,ALT,LDH,ALP,GGT) to check the drug-related safety in 10 lung cancer patients on POD 1 (IU/L)
Clinical chemistry examination-12 | postoperative day 5
  Carrying out the clinical chemistry examination (AST,ALT,LDH,ALP,GGT) to check the drug-related safety in 10 lung cancer patients on POD 5 (IU/L)
Clinical chemistry examination-13 | within two weeks before surgery
  Carrying out the clinical chemistry examination (Na, K, Cl) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (mmol/L)
Clinical chemistry examination-14 | postoperative day 0
  Carrying out the clinical chemistry examination (Na, K, Cl) to check the drug-related safety in 10 lung cancer patients on POD 0 (mmol/L)
Clinical chemistry examination-15 | postoperative day 1
  Carrying out the clinical chemistry examination (Na, K, Cl) to check the drug-related safety in 10 lung cancer patients on POD 1 (mmol/L)
Clinical chemistry examination-16 | postoperative day 5
  Carrying out the clinical chemistry examination (Na, K, Cl) to check the drug-related safety in 10 lung cancer patients on POD 5 (mmol/L)
Hematology examination-1 | within two weeks before surgery
  Carrying out the clinical chemistry examination (Mg) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery(mEq/L)
Hematology examination-2 | postoperative day 0
  Carrying out the clinical chemistry examination (Mg) to check the drug-related safety in 10 lung cancer patients on POD 0 (mEq/L)
Hematology examination-3 | postoperative day 1
  Carrying out the clinical chemistry examination (Mg) to check the drug-related safety in 10 lung cancer patients on POD 1 (mEq/L)
Hematology examination-4 | postoperative day 5
  Carrying out the clinical chemistry examination (Mg) to check the drug-related safety in 10 lung cancer patients on POD 5 (mEq/L)
Hematology examination-5 | within two weeks before surgery
  Carrying out the clinical hematology examination (hemoglobin, MCHC) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (g/dL)
Hematology examination-6 | postoperative day 0
  Carrying out the clinical hematology examination (hemoglobin, MCHC) to check the drug-related safety in 10 lung cancer patients on POD 0 (g/dL)
Hematology examination-7 | postoperative day 1
  Carrying out the clinical hematology examination (hemoglobin, MCHC) to check the drug-related safety in 10 lung cancer patients on POD 1 (g/dL)
Hematology examination-8 | postoperative day 5
  Carrying out the clinical hematology examination (hemoglobin, MCHC) to check the drug-related safety in 10 lung cancer patients on POD 5 (g/dL)
Hematology examination-9 | within two weeks before surgery
  Carrying out the clinical hematology examination (hematocrit, WBC differential) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (%)
Hematology examination-10 | postoperative day 0
  Carrying out the clinical hematology examination (hematocrit, WBC differential) to check the drug-related safety in 10 lung cancer patients on POD0 (%)
Hematology examination-11 | postoperative day 1
  Carrying out the clinical hematology examination (hematocrit, WBC differential) to check the drug-related safety in 10 lung cancer patients on POD1 (%)
Hematology examination-12 | postoperative day 5
  Carrying out the clinical hematology examination (hematocrit, WBC differential) to check the drug-related safety in 10 lung cancer patients on POD5 (%)
Hematology examination-13 | within two weeks before surgery
  Carrying out the clinical hematology examination (RBC count, WBC count, platelet count) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (10³/μl)
Hematology examination-14 | postoperative day 0
  Carrying out the clinical hematology examination (RBC count, WBC count, platelet count) to check the drug-related safety in 10 lung cancer patients on POD0 (10³/μl)
Hematology examination-15 | postoperative day 1
  Carrying out the clinical hematology examination (RBC count, WBC count, platelet count) to check the drug-related safety in 10 lung cancer patients on POD1 (10³/μl)
Hematology examination-16 | postoperative day 5
  Carrying out the clinical hematology examination (RBC count, WBC count, platelet count) to check the drug-related safety in 10 lung cancer patients on POD5 (10³/μl)
Hematology examination-17 | within two weeks before surgery
  Carrying out the clinical hematology examination (MCV) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery(fL)
Hematology examination-18 | postoperative day 0
  Carrying out the clinical hematology examination (MCV) to check the drug-related safety in 10 lung cancer patients on POD 0 (fL)
Hematology examination-19 | postoperative day 1
  Carrying out the clinical hematology examination (MCV) to check the drug-related safety in 10 lung cancer patients on POD 1(fL)
Hematology examination-20 | postoperative day 5
  Carrying out the clinical hematology examination (MCV) to check the drug-related safety in 10 lung cancer patients on POD 5 (fL)
Hematology examination- 21 | within two weeks before surgery
  Carrying out the clinical hematology examination (MCH) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (pg)
Hematology examination- 22 | postoperative day 0
  Carrying out the clinical hematology examination (MCH) to check the drug-related safety in 10 lung cancer patients and POD 0 (pg)
Hematology examination- 23 | postoperative day 1
  Carrying out the clinical hematology examination (MCH) to check the drug-related safety in 10 lung cancer patients on POD 1 (pg)
Hematology examination- 24 | postoperative day 5
  Carrying out the clinical hematology examination (MCH) to check the drug-related safety in 10 lung cancer patients on POD 5 (pg)
Hematology examination- 25 | within two weeks before surgery
  Carrying out the clinical hematology examination (PT, aPTT) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (sec)
Hematology examination- 26 | postoperative day 0
  Carrying out the clinical hematology examination (PT, aPTT) to check the drug-related safety in 10 lung cancer patients on POD 0 (sec)
Hematology examination- 27 | postoperative day 1
  Carrying out the clinical hematology examination (PT, aPTT) to check the drug-related safety in 10 lung cancer patients on POD 1 (sec)
Hematology examination- 28 | postoperative day 5
  Carrying out the clinical hematology examination (PT, aPTT) to check the drug-related safety in 10 lung cancer patients on POD 5 (sec)
Check for changes of urinalysis-1 | within two weeks before surgery
  Carrying out the urinalysis examination(specific gravity, pH, glucose, bilirubin in urine) within two weeks before surgery (number)
Check for changes of urinalysis-2 | postoperative day 0
  Carrying out the urinalysis examination(specific gravity, pH, glucose, bilirubin in urine) on POD 0 (number)
Check for changes of urinalysis-3 | postoperative day 1
  Carrying out the urinalysis examination(specific gravity, pH, glucose, bilirubin in urine) on POD 1(number)
Check for changes of urinalysis-4 | postoperative day 5
  Carrying out the urinalysis examination(specific gravity, pH, glucose, bilirubin in urine) on POD 5 (number)
Check for changes of urinalysis-5 | within two weeks before surgery
  Carrying out the urinalysis examination(ketone, blood, protein, urobilinogen, nitrate in urine) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery (0 or +1)
Check for changes of urinalysis-6 | postoperative day 0
  Carrying out the urinalysis examination(ketone, blood, protein, urobilinogen, nitrate in urine) to check the drug-related safety in 10 lung cancer patients on POD 0 (0 or +1)
Check for changes of urinalysis-7 | postoperative day 1
  Carrying out the urinalysis examination(ketone, blood, protein, urobilinogen, nitrate in urine) to check the drug-related safety in 10 lung cancer patients on POD 1 (0 or +1)
Check for changes of urinalysis-8 | postoperative day 5
  Carrying out the urinalysis examination(ketone, blood, protein, urobilinogen, nitrate in urine) to check the drug-related safety in 10 lung cancer patients on POD 5 (0 or +1)
Check for changes of urinalysis-9 | within two weeks before surgery
  Carrying out the urinalysis examination(WBC in urine) to check the drug-related safety in 10 lung cancer patients within two weeks before surgery(4 - 0 / HPF
Check for changes of urinalysis-10 | postoperative day 0
  Carrying out the urinalysis examination(WBC in urine) to check the drug-related safety in 10 lung cancer patients on POD 0 (4 - 0 / HPF)
Check for changes of urinalysis-11 | postoperative day 1
  Carrying out the urinalysis examination(WBC in urine) to check the drug-related safety in 10 lung cancer patients on POD 1 (4 - 0 / HPF)
Check for changes of urinalysis-12 | postoperative day 5
  Carrying out the urinalysis examination(WBC in urine) to check the drug-related safety in 10 lung cancer patients on POD 5 (4 - 0 / HPF)
Observation of the irritable adverse reaction | Up to 2 hours after drug injection
  Observation of the irritable adverse reaction (Urticaria, angioedema, allergic rhinitis, anaphylaxis, exanthermatous eruption, fixed drug eruption, acneiform eruption, purpura eruption, urticarial eruption, bullous eruption, lichenoid eruption, Stevens-Johnson syndrom, acute generalized exanthematous pustulosis, toxic epidermal necrolysis) to check the drug-related safety in 10 lung cancer patients
Effective dose measurement | Up to five days after surgery

SECONDARY OUTCOMES:
Confirm the sentinel lymph node identification rate | Through study completion, an average of 1 year
  Calculation the percentage of cancer cells found in pathological test among sentinel lymph nodes where fluorescent or nuclear signal are detected.
Confirm the false negative rate | Through study completion, an average of 1 year
  Calculation the proportion of cancer cells found in pathological tests among non-sentinel lymph nodes where no fluorescent or nuclear signals were detected.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Koo Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No